CLINICAL TRIAL: NCT04059575
Title: What Kind of Kinesio Taping Material Should be Used to Decrease the Injury Risk Better
Brief Title: Is Kinesio Taping Application Effective on Decreasing Injury Risk for Tennis Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guven Health Group (Other)
Collaborators: Hacettepe University (Other); Baskent University (Other)
Responsible Party: Principal Investigator, GUL BALTACI, PROFESSOR, PT, PH.D, Guven Health Group
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 511
Record Dates: First submitted 2019-07-24; First posted 2019-08-16 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Injury
Keywords: tennis; vertical jump; kinesio taping; thermography
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The part of muscle with more activation (greater heat) was measured by the thermo graphic camera and the heat was recorded in centigrade. Each participant was thermo graphically evaluated in the same room (ambient temperature, 21°C) and participants were left for 10-20 minutes to 'acclimatize' to the thermographic imaging environment FLIR E5 Thermal Camera, with a resolution of 120 x 90 pixels was used for thermal imaging and the Color Palette iron was chosen for displaying the images. It is indicated that IR imaging may be a reliable and valid measure of treatment outcomes with clinical utility and sensitivity
Who Masked: Participant
Masking Description: Thirty-three young tennis players aged between 9 and 12 yrs were recruited in the study. The exclusion criteria included those (a) with soft tissue or bone problems affecting lower extremity, (b) who had acute inflammation affecting lower extremity region, (c) had scoliosis, (d) who had undergone any orthopedic surgery, (e) who had defined any pain or painful area at lower extremities and (f) who were obese (BMI>30 kg/m2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PERFORMANCE PLUS (Experimental): performance plus better than GOLD TEX
  Interventions: Other: Kinesio Taping (Performance Plus)
- GOLD TEX (Active Comparator): GOLD TEX better than performance plus
  Interventions: Other: Kinesio taping (Gold Tex)

INTERVENTIONS:
Other: Kinesio Taping (Performance Plus) — PP and GT taping applications were done by using kinesio taping muscle facilitation techniques to Quadriceps and Gastrosoleus muscles. I tape with a tension of 10-35% was used for muscle facilitation. All patients were assessed by an experienced physiotherapist, and the tapings were done by another experienced physiotherapist in order to provide a single blind structure of the study.
  Arms: PERFORMANCE PLUS
Other: Kinesio taping (Gold Tex) — PP and GT taping applications were done by using kinesio taping muscle facilitation techniques to Quadriceps and Gastrosoleus muscles. I tape with a tension of 10-35% was used for muscle facilitation. All patients were assessed by an experienced physiotherapist, and the tapings were done by another experienced physiotherapist in order to provide a single blind structure of the study.
  Arms: GOLD TEX

SUMMARY:
Research design: The study protocol was approved and required permissions were taken from related tennis club officials, and a written consent was obtained from all the participants' parents about the study. Thirty-three young tennis players aged between 9 and 12 were included in our study. Assessment were done bare (no tape), after 45 min of performance plus kinesio taping application (PP application) and after 45 min of gold text FP kinesio taping application (GT application). We were randomly taped with either PP or GT taping applications using an online random allocation software program (GraphPad Software QuickCalcs, GraphPad Software Inc., La Jolla, CA, USA). Thirty min of rest was given between 2 taping applications after the removal of the first tape. One participant was not able to complete the second taping procedure. PP and GT taping applications were done by using kinesio taping muscle facilitation techniques to Quadriceps and Gastrosoleus muscles. I-shaped tape with a tension of 10-35% was used for muscle facilitation. All patients were assessed by an experienced physiotherapist, and the tapings were done by another experienced physiotherapist in order to provide a single blind structure of the study.

DETAILED DESCRIPTION:
Participants: Thirty-three young tennis players aged between 9 and 12 yrs were recruited in the study. The exclusion criteria included those (a) with soft tissue or bone problems affecting lower extremity, (b) who had acute inflammation affecting lower extremity region, (c) had scoliosis, (d) who had undergone any orthopedic surgery, (e) who had defined any pain or painful area at lower extremities and (f) who were obese (BMI>30 kg/m2).

Assessments: Thermal analysis was done for risk of injury including both lower extremities. Quadriceps muscle was chosen from upper leg and gastro soleus muscle was chosen from lower leg region for thermal analysis. The thermo graphic assessment was performed by using FLIR E5 (FLIR Systems AB, Sweden) thermal camera in order to evaluate which muscles had the highest thermal activity while maintaining stable upright posture. The part of muscle with more activation (greater heat) was measured by the thermo graphic camera and the heat was recorded in centigrade. Each participant was thermo graphically evaluated in the same room (ambient temperature, 21°C) and participants were left for 10-20 minutes to 'acclimatize' to the thermographic imaging environment FLIR E5 Thermal Camera, with a resolution of 120 x 90 pixels was used for thermal imaging and the Color Palette iron was chosen for displaying the images. It is indicated that IR imaging may be a reliable and valid measure of treatment outcomes with clinical utility and sensitivity

The power analysis indicated that 33 participants for total were needed with 80 % power and a 5 % type 1 error. The power analysis of our study showed a power of 80% with tissue temperature as the primary outcome. The data were analyzed using statistical software (SPSS version 18, Inc., Chicago, IL, USA). All the statistical analyses were set a priori at an alpha level of p<0.05. The tests for homogeneity (Levene's test) and normality (Shapiro-Wilk) were used to determine the appropriate statistical methods. According to the test results, nonparametric Friedman test was used for comparisons between baseline, first taping and last taping. Wilcoxon test was used for possible differences which may occur between taping applications in order to identify the application that provided the difference. Parametric test assumptions were not possible due to small sample size and inhomogeneous parameters.

ELIGIBILITY:
Inclusion Criteria:

* at least playing tennis 2 years
* to be between 9 and 12 years
* no any sport activity-only tennis
* to be a volunteer

Exclusion Criteria:

1. with soft tissue or bone problems affecting lower extremity,
2. who had acute inflammation affecting lower extremity region,
3. had scoliosis,
4. who had undergone any orthopedic surgery,
5. who had defined any pain or painful area at lower extremities and
6. who were obese (BMI>30 kg/m2).

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
termal analysis | 2 hours
  Quadriceps muscle was chosen from upper leg and gastro soleus muscle was chosen from lower leg region for thermal analysis. The thermo graphic assessment was performed by using FLIR E5 (FLIR Systems AB, Sweden) thermal camera in order to evaluate which muscles had the highest thermal activity while maintaining stable upright posture. The part of muscle with more activation (greater heat) was measured by the thermo graphic camera and the heat was recorded in centigrade. Each participant was thermo graphically evaluated in the same room (ambient temperature, 21°C) and participants were left for 10-20 minutes to 'acclimatize' to the thermographic imaging environment FLIR E5 Thermal Camera, with a resolution of 120 x 90 pixels was used for thermal imaging.
vertical jump | 1 hours
  A vertical jump test was performed before and after the application of Kinesio taping® to their quadriceps and gastrocnemius muscles according to Kase's recommendations. The height and flight time data was collected using a portable optical timing system (Optojump Next; Microgate, Bolzano, Italy) during a counter movement jump. Mean maximum jump height and flight time were averaged from three attempts. Two-way repeated measures ANOVAs were used to assess the influence taping condition on vertical jump performance.

SECONDARY OUTCOMES:
age | through study completion, an average of 8 weeks
  Sports age is important to determine the description of differences between ages and sexes.

CONTACTS AND LOCATIONS:
Overall Officials: YESIM S CETINKAYA, MD, Study Director — Guven Health Group
Locations (1):
- Guven Health Group, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Each participant was thermo graphically evaluated in the same room (ambient temperature, 21°C) and participants were left for 10-20 minutes to 'acclimatize' to the thermographic imaging environment FLIR E5 Thermal Camera, with a resolution of 120 x 90 pixels was used for thermal imaging and the Color Palette iron was chosen for displaying the images. It is indicated that IR imaging may be a reliable and valid measure of treatment outcomes with clinical utility and sensitivity

REFERENCES:
- [Result] Bicici S, Karatas N, Baltaci G. Effect of athletic taping and kinesiotaping(R) on measurements of functional performance in basketball players with chronic inversion ankle sprains. Int J Sports Phys Ther. 2012 Apr;7(2):154-66. PMID 22530190
- [Result] Kirmizigil B, Chauchat JR, Yalciner O, Iyigun G, Angin E, Baltaci G. The Effectiveness of Kinesio Taping in Recovering From Delayed Onset Muscle Soreness: A Crossover Study. J Sport Rehabil. 2019 Oct 18;29(4):385-393. doi: 10.1123/jsr.2018-0389. Print 2020 May 1. PMID 30860409
- [Result] Thomas MG, Mohan D, Sahasi G, Prabhu GG. Personality and attitude correlates of drug abuse amongst students of a high school in Delhi: a replicated study. Indian J Med Res. 1979 Jun;69:990-5. No abstract available. PMID 468356
- See also: Kinesiotaping related articles — http://www.kinesiotaping.com